CLINICAL TRIAL: NCT01877356
Title: Unilateral Versus Bilateral Spinal Anesthesia in Day Case Procedures: Difference in Block Characteristics, Micturition Quality and Discharge Time
Brief Title: Comparative Study Between Bilateral and Unilateral Spinal Anaesthesia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: intermittent evaluation of results: high incendence of complications
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Dr M. B. Breebaart, dr, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: study B300201215548; B300-2012-15-548 (Other: BUN (belgisch uniek nummer))
Record Dates: First submitted 2013-03-29; First posted 2013-06-13 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Anesthesia; Adverse Effect, Spinal and Epidural
Keywords: ambulatory surgery; spinal anesthesia; micturition; bladder retention; unilateral block; prilocaine hyperbaric; prilocaine plain; local anaesthetic dose
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bilateral spinal anesthesia (Experimental): bilateral spinal anesthesia prilocaine plain 20% 50 mg ambulatory surgery
  Interventions: Procedure: bilateral spinal anesthesia
- unilateral spinal anesthesia (Experimental): unilateral spinal anesthesia prilocaine hyperbaar 2% 30 mg ambulatory surgery
  Interventions: Procedure: unilateral spinal anesthesia

INTERVENTIONS:
Procedure: bilateral spinal anesthesia — prilocaine plain 2% 50 mg
  Arms: bilateral spinal anesthesia
Procedure: unilateral spinal anesthesia — prilocaine 2% hyperbaric 30 mg
  Arms: unilateral spinal anesthesia

SUMMARY:
The purpose of this study is to compare unilateral spinal anesthesia using hyperbaric Prilocaine with "classical bilateral spinal anesthesia" using plain Prilocaine according to block characteristics and quality of micturition, standardized to the subjects own functional bladder capacity. Our hypothesis is that unilateral spinal anesthesia will provide faster time to micturtition and discharge, lesser hypotension and lesser micturition problems.

DETAILED DESCRIPTION:
Many studies have been published in search of the ideal locoregional anesthetic for day case procedures under spinal anesthesia.

Transient neurological symptoms (TNS) and bladder retention are two side effects, which have been described in literature with incidences ranging from 0-80%.

Lidocaine, which was our hospital standard for spinal anesthesia in day case surgery, has a high incidence of TNS. Besides changing the product, dose or additive, optimisation of spinal anesthesia can be performed by changing anesthetic technique or fluid policy.

There is no consensus in literature about fluid policy and the risk of urinary retention. In a previous study we found that urge sensation and bladder capacity is subject to a high variability.

There are a few studies published about unilateral anesthesia for day-case surgery. For bilateral anesthesia it was shown that recuperation of the detrusor function comes with the regression of the sensory block to the S2 dermatome . However, little is known about bladder function during unilateral block of the sacral segments, not to mention the detrusor function and micturition with an asymmetric recovery of the sensory and motor block.

Prilocaine has found to induce reasonably short durations of spinal blockade, without causing TNS while manufactured in plain and hyperbaric solutions .

We expect that with a unilateral technique patients can void faster and can reach discharge criteria faster then with a bilateral technique.

We will compare unilateral spinal anesthesia with hyperbaric prilocaine with bilateral spinal anesthesia with plain prilocaine. The two techniques will be compared on the following subject

* quality of the motor and sensory block
* recovery from the sensory and motor block
* hemoynamic changens (blood pressure and hart rate)
* time to micturition
* micturition quality
* discharge time
* complications

Sensory block will be tested by loss of cold sensation. Quality of unilateral block will be tested by QST.

Protocol for catheterisation will be adjusted according to the patients individual bladder capacitity, based on a bladder diary. Quality of micturition will be based on bladderscanning, uroflow and subjective complaints. A micturition score from one of our previous studies is used.

Two days and one week postoperative patients will be called and asked if they experienced one of the following symptoms:

* Back pain
* Symptoms of TNS
* Headache
* Micturition problems
* Use of per oral pain medication
* Other

ELIGIBILITY:
Inclusion Criteria:

* spinal anaesthesia
* surgery<60 minutes

Exclusion Criteria:

* preexisting micturition problems
* surgery lower abdomen/pelvis
* bmi>30
* mental problems
* kidney disease
* neurologic disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2012-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
time to micturition (minutes) | up to 360 minutes
  time to event outcome. Time from injection untill patient the moment voids for the first time (average off 4hours)
discharge time ( minutes) | up to 360 minutes
  time from injection untill dischargecriteria are reached ( average of 4 hours). Time to event outcome , event = discharge
regression motor block | up to 240 minutes
  Motor block will be assessed at regular intervals from spinal injection (t0) until total regression of the motor block.

SECONDARY OUTCOMES:
drop blood pressure | up to 240 minutes
  percentage drop blood pressure compared to baseline ( measured before spinal injection) Blood pressure will be measured at regular intervals from just prior to spinal injection until discharge
incidence transient neurologic symptoms | 1 week
  patients will be called at home one week postoperatively to ask for symptoms resembling transien neurological symptoms

CONTACTS AND LOCATIONS:
Overall Officials: margaretha breebaart, md, Principal Investigator — senior member of staff department anaesthesiology; Marcel Vercauteren, professor, Study Director — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

REFERENCES:
- [Background] Esmaoglu A, Karaoglu S, Mizrak A, Boyaci A. Bilateral vs. unilateral spinal anesthesia for outpatient knee arthroscopies. Knee Surg Sports Traumatol Arthrosc. 2004 Mar;12(2):155-8. doi: 10.1007/s00167-003-0350-2. Epub 2003 Feb 22. PMID 15024563
- [Background] Fanelli G, Borghi B, Casati A, Bertini L, Montebugnoli M, Torri G. Unilateral bupivacaine spinal anesthesia for outpatient knee arthroscopy. Italian Study Group on Unilateral Spinal Anesthesia. Can J Anaesth. 2000 Aug;47(8):746-51. doi: 10.1007/BF03019476. PMID 10958090
- [Background] Akhtar MN, Tariq S, Abbas N, Murtaza G, Nadeem Naqvi SM. Comparison of haemodynamic changes in patients undergoing unilateral and bilateral spinal anaesthesia. J Coll Physicians Surg Pak. 2012 Dec;22(12):747-50. PMID 23217477
- [Background] Choi S, Mahon P, Awad IT. Neuraxial anesthesia and bladder dysfunction in the perioperative period: a systematic review. Can J Anaesth. 2012 Jul;59(7):681-703. doi: 10.1007/s12630-012-9717-5. Epub 2012 Apr 26. PMID 22535232
- [Background] Kamphuis ET, Ionescu TI, Kuipers PW, de Gier J, van Venrooij GE, Boon TA. Recovery of storage and emptying functions of the urinary bladder after spinal anesthesia with lidocaine and with bupivacaine in men. Anesthesiology. 1998 Feb;88(2):310-6. doi: 10.1097/00000542-199802000-00007. PMID 9477049
- [Background] Breebaart MB, Vercauteren MP, Hoffmann VL, Adriaensen HA. Urinary bladder scanning after day-case arthroscopy under spinal anaesthesia: comparison between lidocaine, ropivacaine, and levobupivacaine. Br J Anaesth. 2003 Mar;90(3):309-13. doi: 10.1093/bja/aeg078. PMID 12594142